CLINICAL TRIAL: NCT05618119
Title: The Impact of Gender Differences in P-glycoprotein Function Measured With [18F]MC225 and PET
Brief Title: [18F]MC225 PET to Evaluate Gender Differences in BBB P-gp Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Gert Luurtsema, Prof., University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11323
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Gender
Keywords: P-glycoprotein; MC225; [18F]MC225; PET
MeSH Terms: conditions — Coitus | interventions — MC225 compound

STUDY DESIGN:
Intervention Model Description: Two groups of healthy volunteers (5 male, 5 female)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male (Active Comparator): 5 male participants will undergo a [18F]MC225 PET scan
  Interventions: Drug: [18F]MC225
- Female (Active Comparator): 5 female participants will undergo a [18F]MC225 PET scan
  Interventions: Drug: [18F]MC225

INTERVENTIONS:
Drug: [18F]MC225 — [18F]MC225 PET scan

SUMMARY:
P-gp is one of the main efflux transporters at the blood-brain barrier and is responsible for the transport of a variety of neurotoxic substances, including pharmaceuticals. Multiple studies report gender differences in therapeutic outcomes, toxicity and side effects for many drug agents. P-gp plays an important role in the bio-availability, drug distribution, metabolism and elimination of pharmaceuticals labelled as P-gp substrates (e.g. the majority of antidepressants and antipsychotics). A difference in P-gp function was already reported in hepatic P-gp expression. The aim of the current study is to evaluate the influence of gender on cerebral P-gp function. Outcomes of this study can be of great importance in gender-based prescription of P-gp substrate pharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Use of medication with a known effect on the BBB P-glycoprotein transporter
* Any history of neurological or psychiatric conditions affecting the BBB P-glycoprotein function

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
PET kinetic modeling outcome parameters [18F]MC225 | 60 minutes after administration [18F]MC225
  volume of distribution, K1, k2

SECONDARY OUTCOMES:
PET kinetic modeling outcome parameters [15O]H2O | 10 minutes after administration of [15O]H2O
  K1 to evaluate Cerebral Blood Flow (CBF)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salvi de Souza G, Mossel P, Somsen JF, Providencia L, Bartels AL, Willemsen ATM, Dierckx RAJO, Furini CRG, Lammertsma AA, Tsoumpas C, Luurtsema G. Evaluating image-derived input functions for cerebral [18F]MC225 PET studies. Front Nucl Med. 2025 Jun 5;5:1597902. doi: 10.3389/fnume.2025.1597902. eCollection 2025. PMID 40538986